CLINICAL TRIAL: NCT01388855
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Vitamin D in Heart Failure: A Pilot Study
Brief Title: Pilot Study of Vitamin D Supplementation in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Responsible Party: Principal Investigator, Liz, Clinical Resource Dietitian, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011-028
Record Dates: First submitted 2011-06-22; First posted 2011-07-07 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure
Keywords: Heart Failure; Vitamin D; Pain; Pilot Study; RCT
MeSH Terms: conditions — Heart Failure; Pain | interventions — Cholecalciferol; Vitamin D; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecalciferol (Experimental): Patients were given two cholecalciferol tablets (10,000 IU each) daily for 30 days.
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): Patients were given two cholecalciferol placebo tablets daily for 30 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Subjects receive cholecalciferol 20,000 IU daily for 30 days followed by 20,000 IU once weekly for 8 weeks.
  Other Names: Vitamin D
  Arms: Cholecalciferol
Drug: Placebo — Pills made to look like vitamin D but have no medication in them
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the methods are feasible for a larger clinical trial.The study will examine the relationship between vitamin D status, quality of life, pain and walking distance of individuals living with heart failure.

DETAILED DESCRIPTION:
This study is being conducted as a pilot project to determine the feasibility of the methods to inform the conduct of a future larger study. This double-blind randomized controlled trial will examine the relationship between vitamin D status, Quality of Life (QOL), pain and functional capacity of individuals living with heart failure (HF) pre and post vitamin D supplementation. The study outcome measures include: the rate of recruitment, retention and compliance with the study procedures. Quality of life will be measured by the EQ-5D™ questionnaire; the Brief Pain Inventory (BPI) will be used to evaluate subject pain. The 6-minute walk test (6MWT) will evaluate functional capacity. Serum 25-hydroxyvitamin D (25OHD) levels will quantify the adequacy of vitamin D dosing to achieve target 25OHD levels.

A convenience sample of 40 subjects (20 per treatment group) will be prospectively recruited from the Royal Columbian Hospital (RCH) Heart Function (HFx) Clinic. Subjects will be randomized to receive either vitamin D3 (cholecalciferol) or a matching placebo at a dose of 20,000 IU daily for 30 days followed by 20,000 IU once weekly for 8 weeks. Subjects will have their 25OHD levels measured, self-administer the EQ-5D™ and BPI questionnaires and perform the 6MWT at the study entry and again at the completion of the study (12 weeks after entry).

Descriptive statistics (mean, standard deviation and proportion as appropriate) will be used to describe the data. The feasibility of all study procedures will be reported by percentage and compared to the standard set by the team of 80%.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* New York Heart Association functional Class II or III symptoms
* Ability to communicate in English or through a translator
* Competent to sign the informed consent

Exclusion Criteria:

* Co-morbidity that would negatively impact quality of life (e.g. severe arthritis, or fibromyalgia)
* Co-morbidity that would negatively impact vitamin D metabolism (glomerular filtration rate-15-29%, significant liver dysfunction
* On a pharmaceutical agent that could lower Vitamin D levels (e.g. glucocorticoids, anticonvulsants)
* Taking >600 IU vitamin D (cholecalciferol or ergocalciferol) daily
* Moderate or severe cognitive impairment
* Contraindication to vitamin D supplementation: history of hypercalcemia or conditions that increase the risk of hypercalcemia (sarcoidosis, tuberculosis or lymphoma)
* Wheelchair bound (ambulation is a component of the QOL questionnaire

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Rate of participant recruitment | 6 months
  The percentage of patients recruited from those that present to clinic.
Participant compliance with study procedures | 6 months
  Proportion completing the quality of life questionnaire, 6 minute walk test and medication regimen
Participant rate of retention | 6 months
  Proportion of participants retained in study

SECONDARY OUTCOMES:
Number of participants with hypercalcemia as a measure of safety and tolerability. | 6 months
Number of participants that achieve a target serum 25-hydroxyvitamin D of 75nmol/L | 8 months
The values achieved for quality of life and pain questionnaire and functional capacity measure. | 8 months
  Quality of life will be measured by the EQ-5D questionnaire. Pain will be measured by the Brief Pain Inventory questionnaire. Functional capacity will be measured by the standardized and validated 6 minute walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Liz C da Silva, MS, Principal Investigator — Fraser Health Authority
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada